CLINICAL TRIAL: NCT04473807
Title: Feasibility and Safety of Intravenous Sotalol Administered as a Loading Dose to Initiate Oral Sotalol Therapy in Adult Patients With Atrial Fibrillation (DASH-AF)
Brief Title: Feasibility and Safety of IV Sotalol Administered as a Loading Dose to Initiate Oral Sotalol Therapy
Acronym: DASH-AF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Texas Cardiac Arrhythmia Research Foundation (Other); Munson Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KCHRF-DASH-AF-0002
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-02

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation
Keywords: Sotalol, Intravenous, Oral, Arrhythmias, Atrial Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DASH-AF (Other): Patients with history of highly symptomatic persistent or paroxysmal AF who are scheduled for sotalol therapy once in sinus rhythm will be enrolled in this study.
  Interventions: Drug: Intravenous Sotalol Administered as a Loading Dose to Initiate Oral Sotalol Therapy in Adult Patients with Atrial Fibrillation

INTERVENTIONS:
Drug: Intravenous Sotalol Administered as a Loading Dose to Initiate Oral Sotalol Therapy in Adult Patients with Atrial Fibrillation — The hypothesis to be tested is that the intravenous loading regimen followed by oral sotalol administration 4 hours after the conclusion of the IV infusion (every 12 hours thereafter) will result in sotalol peak concentrations at the end of IV loading dose (IV to oral loading) which are comparable to the steady state and maximum QTc seen on Day 3 after the last in-hospital oral dose.
  Other Names: Intravenous Sotalol Administered as a Loading Dose to Initiate Oral Sotalol Therapy

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the IV loading strategy in patients who are selected to receive sotalol.

DETAILED DESCRIPTION:
This is an open-label single arm study investigating the safety and feasibility of an intravenous loading regimen of sotalol to initiate patients on oral sotalol therapy. Informed Consent will be obtained from all patients prior to enrollment in the study. Patients will be admitted to the hospital in accordance with standard hospital protocol for oral sotalol loading.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 18 - 85 years old
* Recent (within 1 day) cardioversion for atrial fibrillation with scheduled sotalol therapy
* History of highly symptomatic atrial fibrillation who are scheduled for sotalol therapy
* Creatinine clearance ≥60 mL/min
* Subject has provided informed consent prior to initiation of any study-specific activities/procedures

Exclusion Criteria:

* Baseline bradycardia (<50 bpm) off all antiarrhythmic drugs and or Atrioventricular nodal blocking drugs
* Sick sinus syndrome, unless a functioning pacemaker is present.
* Any known sensitivities to beta-blockers
* Uncontrolled heart failure
* Second-degree (Mobitz II, Wenckebach) or third-degree atrioventricular block
* Recent (within 7 days) surgical or catheter ablation procedure
* Severe electrolyte abnormalities (including serum K<3.5)
* Known use of other QTc prolonging drugs (See Appendix A)
* Recent (within 7 days) sotalol use
* Baseline QTc >450 ms
* Severe reactive airway disease - defined as difficulty breathing from bronchial tubes, swelling and overreaction to an irritant
* History of Torsade de Pointes (TdP)
* Pregnancy or breastfeeding
* Left ventricular ejection fraction (LVEF) less than 35%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
intravenous loading regimen followed by q12h oral sotalol administration | 3 months
  The hypothesis to be tested is that the intravenous loading regimen followed by q12h oral sotalol administration will result in sotalol concentration and QTc peaks on day 1 (IV to oral loading) which are comparable to the steady-state and maximum QTc seen on Day 3 (steady-state).

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Research Foundation
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boriani G, Valzania C, Biffi M, Corazza I, Camanini C, Martignani C, Bacchi L, Zannoli R, Branzi A. Increase in QT/QTc dispersion after low energy cardioversion of chronic persistent atrial fibrillation. Int J Cardiol. 2004 Jun;95(2-3):245-50. doi: 10.1016/j.ijcard.2003.05.022. PMID 15193827
- [Background] Darbar D, Hardin B, Harris P, Roden DM. A rate-independent method of assessing QT-RR slope following conversion of atrial fibrillation. J Cardiovasc Electrophysiol. 2007 Jun;18(6):636-41. doi: 10.1111/j.1540-8167.2007.00817.x. Epub 2007 May 3. PMID 17488270
- [Background] HIGHLIGHTS OF PRESCRIBING INFORMATION: Sotalol hydrochloride injection for intravenous use. https://www.accessdata.fda.gov/drugsatfda_docs/label/2009/022306s000lbl.pdf.
- [Background] Woosley RL, Heise CW, Tate J, Woosley D, Romero KA, Gallo T. QTdrugs List. https://crediblemeds.org/index.php/?cID=328. Accessed August 28, 2019.
- [Derived] Lakkireddy D, Ahmed A, Atkins D, Bawa D, Garg J, Bush J, Charate R, Bommana S, Pothineni NVK, Kabra R, Darden D, Koreber S, Tummala R, Vasamreddy C, Park P, Mohanty S, Gopinathannair R, Seo BW, Natale A, Kennedy R. Feasibility and Safety of Intravenous Sotalol Loading in Adult Patients With Atrial Fibrillation (DASH-AF). JACC Clin Electrophysiol. 2023 Apr;9(4):555-564. doi: 10.1016/j.jacep.2022.11.026. Epub 2023 Feb 22. PMID 37014289